CLINICAL TRIAL: NCT00878462
Title: A Randomized, Crossover Study Evaluating the Acceptability of Unflavored Asenapine and Raspberry Flavored Asenapine in Stable Subjects With A Psychotic Disorder
Brief Title: An Acceptability Study of Unflavored Asenapine Versus Raspberry Flavored Asenapine in Stable Patients With a Psychotic Disorder (P07010)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P07010; A7501024
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Subjects randomly assigned to this sequence receive in order: Treatment A, C, B, A, C, B. Each treatment was one dose, and each patient received a dose in the morning and evening for 3 consecutive days.
  Interventions: Drug: Asenapine WHITE raspberry flavor (Treatment A); Drug: Asenapine RED raspberry flavor (Treatment B); Drug: Asenapine WHITE UNFLAVORED (Treatment C)
- Sequence 2 (Experimental): Subjects randomly assigned to this sequence receive in order: Treatment A, B, C, A, B, C. Each treatment was one dose, and each patient received a dose in the morning and evening for 3 consecutive days.
  Interventions: Drug: Asenapine WHITE raspberry flavor (Treatment A); Drug: Asenapine RED raspberry flavor (Treatment B); Drug: Asenapine WHITE UNFLAVORED (Treatment C)
- Sequence 3 (Experimental): Subjects randomly assigned to this sequence receive in order: Treatment B, C, A, B, C, A. Each treatment was one dose, and each patient received a dose in the morning and evening for 3 consecutive days.
  Interventions: Drug: Asenapine WHITE raspberry flavor (Treatment A); Drug: Asenapine RED raspberry flavor (Treatment B); Drug: Asenapine WHITE UNFLAVORED (Treatment C)
- Sequence 4 (Experimental): Subjects randomly assigned to this sequence receive in order: Treatment B, A, C, B, A, C. Each treatment was one dose, and each patient received a dose in the morning and evening for 3 consecutive days.
  Interventions: Drug: Asenapine WHITE raspberry flavor (Treatment A); Drug: Asenapine RED raspberry flavor (Treatment B); Drug: Asenapine WHITE UNFLAVORED (Treatment C)
- Sequence 5 (Experimental): Subjects randomly assigned to this sequence receive in order: Treatment C, B, A, C, B, A. Each treatment was one dose, and each patient received a dose in the morning and evening for 3 consecutive days.
  Interventions: Drug: Asenapine WHITE raspberry flavor (Treatment A); Drug: Asenapine RED raspberry flavor (Treatment B); Drug: Asenapine WHITE UNFLAVORED (Treatment C)
- Sequence 6 (Experimental): Subjects randomly assigned to this sequence receive in order: Treatment C, A, B, C, A, B. Each treatment was one dose, and each patient received a dose in the morning and evening for 3 consecutive days.
  Interventions: Drug: Asenapine WHITE raspberry flavor (Treatment A); Drug: Asenapine RED raspberry flavor (Treatment B); Drug: Asenapine WHITE UNFLAVORED (Treatment C)

INTERVENTIONS:
Drug: Asenapine WHITE raspberry flavor (Treatment A) — Asenapine (Org 5222), 5 mg white raspberry flavored as fast dissolving tablets
  Other Names: Saphris; Org 5222; SCH 900274
Drug: Asenapine RED raspberry flavor (Treatment B) — Asenapine (Org 5222), 5 mg red raspberry flavored as fast dissolving tablets
  Other Names: Saphris; Org 5222; SCH 900274
Drug: Asenapine WHITE UNFLAVORED (Treatment C) — Asenapine (Org 5222), 5 mg WHITE UNflavored as fast dissolving tablets
  Other Names: Saphris; Org 5222; SCH 900274

SUMMARY:
This trial was a randomized trial to determine a patient's acceptability of unflavored antipsychotic medication compared to raspberry flavored antipsychotic medication. Patients received 6 total doses of study drug (2 doses of each asenapine formulation) over 3 consecutive days: 2 different formulations each day, 1 in the morning and 1 in the evening. The formulations were: white unflavored, white raspberry flavored, and red raspberry flavored. Patients were given a questionnaire following each dose of study medication (one questionnaire twice per day for 3 days) to measure how acceptable each formulation was.

DETAILED DESCRIPTION:
Study drug was administered according to a random selected sequence schedule with 2 constraints: Subjects did not receive consecutive doses of the same formulation, and each formulation was given once in the morning and once in the evening over the course of the 3-day treatment period.

ELIGIBILITY:
Inclusion Criteria:

* are at least 18 years of age and of legal minimum age for trial participation;
* are a male, or a female who is not of childbearing potential
* are free from an acute exacerbation of psychosis for at least 3 months;
* have a current DSM-IV diagnosis of schizophrenia (paranoid, disorganized, catatonic, or undifferentiated subtype), or schizoaffective disorder; delusional disorder, major depressive disorder, or bipolar disorder, for whom chronic antipsychotic therapy is indicated;
* correctly identify 3 out of 4 basic flavors (bitter, sweet, salty, or sour) on a neutral taste paradigm;
* are receiving oral antipsychotic medication.

Exclusion Criteria:

* an uncontrolled, unstable clinically significant medical condition
* clinically significant abnormal laboratory, vital sign, PE, or ECGs findings at Screening;
* previously experienced NMRB (also known as vasovagal reflex) or sensitivity for fainting;
* a positive serum pregnancy test at screening, or the intention to become pregnant within the next 30 days;
* a history of seizures;
* a history of neuromalignant syndrome;
* a current (past 6 months) substance abuse or dependence according to DSM-IV-TR criteria (excluding nicotine);
* an imminent risk of self-harm or harm to others;
* currently receiving a depot antipsychotic, such as fluphenazine decanoate, haloperidol decanoate, or Risperdal Consta, within at least 1 dosing cycle of Day-5;
* any impairment in taste functioning;
* receiving lithium or topiramate;
* judged by the principal investigator (PI) to be unable to reliably respond to the questionnaire based on clinically significant cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2005-06-29 (Actual); Primary Completion 2005-10-15 (Actual); Study Completion 2005-10-15 (Actual)

PRIMARY OUTCOMES:
The response to the question: "How likely would you be to take this medication for at least 1 year if your doctor continued to prescribe it to you and it worked well?"" | After each dose (morning and evening of days 1 through 3)
The response on the following question: "Considering your total impression of this tablet, like the look, the taste and the feel of the tablet, how acceptable is this tablet to you?" | After each dose (morning and evening of days 1 through 3)

SECONDARY OUTCOMES:
Responses on the following question: "How acceptable was the taste of the tablet?" | After each dose (morning and evening of days 1 through 3)